CLINICAL TRIAL: NCT03078192
Title: Non-Invasive Diagnosis of Pulmonary Vascular Disease Using Inhaled 129Xe Magnetic Resonance Imaging
Acronym: XenonMRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bastiaan Driehuys (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Bastiaan Driehuys, Professor, Duke University Medical Center, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro00079617; HHSN268201700001C (Other: National Heart, Lung, and Blood Institutes)
Record Dates: First submitted 2017-02-24; First posted 2017-03-13 (Actual); Results first posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-01

CONDITIONS: Pulmonary Vascular Disease
Keywords: right heart catheterization for evaluation of PAH or other cardiac or pulmonary disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: This will be a single blinded open label study enrolling volunteers and patients with pure PAH (10 subjects), pure left heart disease (10 subjects) and pure lung disease (10 subjects), 5 CTEPH in Aim 1; followed by a larger cohort of 92 subjects with PAH or other cardiac or pulmonary disease for MRI scans
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor, the radiologist who is reading the imaging will be blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training Set - PVD, Isolated Left Heart Failure, Isolated Lung Disease (Experimental): Patients with Pulmonary Vascular Disease (10 subjects), isolated left sided heart failure (10 subjects), and isolated lung disease(10 subjects) will undergo Xe MRI scans with GE-141, Hyperpolarized 129Xenon gas to develop diagnostic criteria for optimizing the sensitivity and specificity of XeMRI for the diagnosis of PVD
  Interventions: Drug: GE-141, Hyperpolarized 129Xenon gas; Device: MRI
- Test Set - Pulmonary Vascular Disease (Experimental): 92 subjects being evaluated for undergoing right heart catheterization for evaluation of PAH or other cardiac or pulmonary disease for testing of diagnostic accuracy of XeMRI for diagnosis of PVD
  Interventions: Drug: GE-141, Hyperpolarized 129Xenon gas; Device: MRI

INTERVENTIONS:
Drug: GE-141, Hyperpolarized 129Xenon gas — XeMRI scans will provide 3D images of ventilation and gas exchange. Subjects will inhale HP 129Xe from the dose delivery bags. Then the subject will be moved into the scanner and they will undergo basic 1H localizer and anatomical scans. Once localization is complete, subjects will under-go several MRI scans after inhalation of HPXe
  Other Names: Xe MRI
Device: MRI — Perform MRI scans with administration of GE-141, Hyperpolarized 129Xenon

SUMMARY:
This study seeks to deploy several forms of 129Xe MRI contrast as well as emerging conventional proton MRI technqiues for imaging lung structure and perfusion. Specifically, the 129Xe MRI scans will provide 3D images of ventilation and gas exchange, and spectroscopic indices will be evaluated to test gas exchange dynamics with high temporal resolution. The conventional 1H MRI scans will include a free-breathing ultra-short echo time (UTE) scan that provides images similar to that of a CT scan. In addition, to characterize perfusion and vascular dimensions directly, patients will undergo a gadolinium-enhanced perfusion scan.

DETAILED DESCRIPTION:
This study seeks to deploy several forms of 129Xe MRI contrast as well as emerging conventional proton MRI technqiues for imaging lung structure and perfusion. Specifically, the 129Xe MRI scans will provide 3D images of ventilation and gas exchange, and spectroscopic indices will be evaluated to test gas exchange dynamics with high temporal resolution. The conventional 1H MRI scans will include a free-breathing ultra-short echo time (UTE) scan that provides images similar to that of a CT scan. In addition, to characterize perfusion and vascular dimensions directly, patients will undergo a gadolinium-enhanced perfusion scan. The overall aims of the study are as follows:

Aim 1. Perform 129Xe MRI scans in cohorts of patients with PVD, isolated left sided heart failure and isolated lung disease:

1.1 Deploy and optimize 129Xe gas exchange MR spectroscopy and imaging, 129Xe ventilation MRI, structural 1H UTE MRI, and breath-hold 1H perfusion MRI.

1.2 Conduct comprehensive 1H-129Xe MRI in 10 patients with pure pulmonary arterial hypertension (PAH) 1.3 Conduct comprehensive MRI in 10 patients with pure left heart failure 1.4 Conduct comprehensive MRI in 10 patients with pure lung disease but no pulmonary hypertension 1.5 Conduct comprehensive MRI in 5 patients with Chronic thromboembolic pulmonary hypertension (CTEPH) pre and post PTE surgery.

Aim 2. Develop diagnostic criteria for optimizing the sensitivity and specificity of 129Xe MRI for the diagnosis of PVD:

2.1 Develop quantification/scoring methods based on PAH, left heart disease, and lung disease MRI 2.2 Develop reader training materials and train 3 expert readers 2.3 Begin prospective recruitment of 92 patients being evaluated for PAH for MRI scans. These patients may be asked to return for a second scan in the study, at a time no earlier than 48hr after their last xenon dose.

Aim 3. Perform a larger, single-blind study testing the diagnostic accuracy of 129Xe MRI for diagnosis of PVD:

3.1 Trained readers will evaluate 129Xe MRI, while blinded to the subject's disease state and will determine the presence and severity of PVD 3.2 Diagnostic accuracy of 129Xe MRI will be compared to the gold standard of hemodynamic and clinical criteria of PAH

1. For this PFTs are not necessary, so they are ancillary
2. However, they are a standard way to characterize patients for publications, etc, so we would like to get them if we can. Getting them from the medical record is perfectly adequate for this pur-pose.

i. If PFTs are not available from the medical record, they are not so critical as to pre-vent us from enrolling the subject. In publications we will simply acknowledge the realities of COVID for this missing data.

This will be an single-blinded, open-label study enrolling volunteers and patients with pure PAH (10 subjects), pure left heart disease (10 subjects) and pure lung disease (10 subjects) [Aim 1] followed by a larger cohort of 92 subjects being evaluated for PAH [Aim 2]. The investigators plan to consent to 127 subjects.

The sample size calculation is based on testing whether the proposed diagnostic test based on Xe MRI has accuracy comparable to imaging diagnostic procedures in clinical practice, such as mammography. To this end, the investigator proposes to test the hypotheses H0: AUC = 0.72 vs. H1: AUC > 0.85, where area under the curve (AUC) is a summary measure of diagnostic accuracy obtained as the the area under the receiver operating characteristic (ROC) curve which displays the tradeoff between sensitivity and specificity for our proposed Xe MRI based diagnostic test. Here AUC = 0.72 represents a moderately accurate test while AUC = 0.85 represents accuracy comparable to clinical mammography. Based on a one sided, one sample test with variances approximated using the binormal model, the investigator estimates a minimum sample size of 46 normals and 46 with disease will be required to test the above hypotheses at a significance level of 5% with 80% power.

ELIGIBILITY:
Inclusion criteria

1. Outpatients of either gender, age > 18
2. Willing and able to give informed consent and adhere to visit/protocol schedules. (Consent must be given before any study procedures are performed)
3. Women of childbearing potential must have a negative urine pregnancy test. This will be confirmed before participation in this investigational protocol.
4. Either has a diagnosis of PAH, isolated left heart disease or lung disease (chronic obstructive pulmonary disease or interstitial lung disease) or CTEPH using established clinical criteria.
5. Patients undergoing right heart catheterization for evaluation of PAH or other cardiac or pulmonary disease for MRI scans

Exclusion criteria

* Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements
* Conditions that will prohibit MRI scanning (metal in eye, claustrophobia, inability to lie supine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with PAH, CTEPH, left heart disease and lung disease will be recruited using inclusion/exclusion criteria. For the first phase of the study, whether patients are receiving approved therapies, enrolled in clinical trials, or receiving no therapy, all will be eligible for inclusion in this study. For the 2nd phase of the study, patients who have PAH and receiving approved therapies, patients who are being evaluated for PVD or other cardiac/pulmonary diseases will be included in the study.
Groups:
- PVD, Left Heart Disease, Lung Disease: The study team recruited 30 subjects. Patients with Pulmonary Vascular Disease (10 subjects), isolated left-sided heart failure (10 subjects), and isolated lung disease(10 subjects) will undergo Xe MRI scans with GE-141, Hyperpolarized 129Xenon gas to develop diagnostic criteria for optimizing the sensitivity and specificity of XeMRI for the diagnosis of PVD
  GE-141, Hyperpolarized 129Xenon gas: XeMRI scans will provide 3D images of ventilation and gas exchange. Subjects will inhale HP 129Xe from the dose delivery bags. Then the subject will be moved into the scanner and they will undergo basic 1H localizer and anatomical scans. Once localization is complete, subjects will under-go several MRI scans after inhalation of HPXe
  MRI: Perform MRI scans with administration of GE-141, Hyperpolarized 129Xenon
- Pulmonary Vascular Disease: the study team recuited 32 subjects being evaluated for undergoing right heart catheterization for evaluation of PAH or other cardiac or pulmonary disease for testing of diagnostic accuracy of XeMRI for diagnosis of PVD
  GE-141, Hyperpolarized 129Xenon gas: XeMRI scans will provide 3D images of ventilation and gas exchange. Subjects will inhale HP 129Xe from the dose delivery bags. Then the subject will be moved into the scanner and they will undergo basic 1H localizer and anatomical scans. Once localization is complete, subjects will under-go several MRI scans after inhalation of HPXe
  MRI: Perform MRI scans with administration of GE-141, Hyperpolarized 129Xenon
Period: Overall Study
Arm/Group | PVD, Left Heart Disease, Lung Disease | Pulmonary Vascular Disease
Started | 30 | 32
Completed | 28 | 28
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 2 | 1
Not completed — screen failure | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- PVD, Left Heart Disease, Lung Disease: Patients with Pulmonary Vascular Disease (10 subjects), isolated left-sided heart failure (10 subjects), and isolated lung disease(10 subjects) will undergo Xe MRI scans with GE-141, Hyperpolarized 129Xenon gas to develop diagnostic criteria for optimizing the sensitivity and specificity of XeMRI for the diagnosis of PVD
  GE-141, Hyperpolarized 129Xenon gas: XeMRI scans will provide 3D images of ventilation and gas exchange. Subjects will inhale HP 129Xe from the dose delivery bags. Then the subject will be moved into the scanner and they will undergo basic 1H localizer and anatomical scans. Once localization is complete, subjects will under-go several MRI scans after inhalation of HPXe
  MRI: Perform MRI scans with administration of GE-141, Hyperpolarized 129Xenon
- Pulmonary Vascular Disease: 92 subjects being evaluated for undergoing right heart catheterization for evaluation of PAH or other cardiac or pulmonary disease for testing of diagnostic accuracy of XeMRI for diagnosis of PVD
  GE-141, Hyperpolarized 129Xenon gas: XeMRI scans will provide 3D images of ventilation and gas exchange. Subjects will inhale HP 129Xe from the dose delivery bags. Then the subject will be moved into the scanner and they will undergo basic 1H localizer and anatomical scans. Once localization is complete, subjects will under-go several MRI scans after inhalation of HPXe
  MRI: Perform MRI scans with administration of GE-141, Hyperpolarized 129Xenon
- Total: Total of all reporting groups
Arm/Group | PVD, Left Heart Disease, Lung Disease | Pulmonary Vascular Disease | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 21 | 43
  >=65 years | 8 | 11 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 20 | 33
  Male | 17 | 12 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 29 | 31 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 6 | 11
  White | 24 | 23 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Participants Determined to be True Positives for Pulmonary Arterial Hypertension
Description: Determine diagnostic accuracy of XeMRI compared to the gold standard of hemodynamic and clinical criteria of pulmonary arterial hypertension (Hemodynamic criteria: mean pulmonary artery pressure > 20 mmHg, pulmonary arterial wedge pressure ≤ 15 mmHg, and pulmonary vascular resistance ≥ 3 Wood units; Clinical criteria: absence of significant systolic dysfunction (LVEF > 40%) or valvular heart disease (moderate or greater mitral or aortic valve disease); absence of significant obstructive or restrictive lung disease; absence of hypoxemic or hypercarbic respiratory failure; absence of chronic thromboembolic disease; absence of sickle cell anemia or other hemolytic anemias; absence of sarcoidosis).
  We used data from Arm 1 (the training set of patients with known pulmonary vascular disease (PVD), isolated left heart disease and lung disease) to determine thresholds for precapillary pulmonary hypertension used for diagnosis in Arm 2 (the test set of pulmonary vascular disease).
Time Frame: up to 2 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Training Set - PVD, Isolated Left Heart Disease, Lung Disease: The study recruited 30 subjects being evaluated for undergoing right heart catheterization for evaluation of PAH or other cardiac or pulmonary disease for testing of diagnostic accuracy of XeMRI for diagnosis of PVD
  GE-141, Hyperpolarized 129Xenon gas: XeMRI scans will provide 3D images of ventilation and gas exchange. Subjects will inhale HP 129Xe from the dose delivery bags. Then the subject will be moved into the scanner and they will undergo basic 1H localizer and anatomical scans. Once localization is complete, subjects will under-go several MRI scans after inhalation of HPXe
  MRI: Perform MRI scans with administration of GE-141, Hyperpolarized 129Xenon
- Test Set - Pulmonary Vascular Disease: The study recruited 32 subjects being evaluated for undergoing right heart catheterization for evaluation of PAH or other cardiac or pulmonary disease for testing of diagnostic accuracy of XeMRI for diagnosis of PVD
  GE-141, Hyperpolarized 129Xenon gas: XeMRI scans will provide 3D images of ventilation and gas exchange. Subjects will inhale HP 129Xe from the dose delivery bags. Then the subject will be moved into the scanner and they will undergo basic 1H localizer and anatomical scans. Once localization is complete, subjects will under-go several MRI scans after inhalation of HPXe
  MRI: Perform MRI scans with administration of GE-141, Hyperpolarized 129Xenon
Arm/Group | Training Set - PVD, Isolated Left Heart Disease, Lung Disease | Test Set - Pulmonary Vascular Disease
Number analyzed (Participants) | 30 | 32
Participants
  By Right Heart Cath: Pre-capillary pulmonary hypertension | 10 | 15
  By Right Heart Cath: Isolated post-capillary pulmonary hypertension | 10 | 5
  By Right Heart Cath: Combined pre- and post-capillary pulmonary hypertension | 0 | 3
  By Right Heart Cath: Pulmonary hypertension (not pre or post) | 0 | 2
  By Right Heart Cath: No pulmonary hypertension | 10 | 7
  By Xenon MRI scan: Pre-capillary pulmonary hypertension | 10 | 18
  By Xenon MRI scan: Isolated post-capillary pulmonary hypertension | 10 | 8
  By Xenon MRI scan: Combined pre- and post-capillary pulmonary hypertension | 0 | 0
  By Xenon MRI scan: Pulmonary hypertension (not pre or post) | 0 | 0
  By Xenon MRI scan: No pulmonary hypertension | 10 | 6
Statistical Analysis 1: Comparison: Training Set - PVD, Isolated Left Heart Disease, Lung Disease; Test type: Other — Detecting pre-capillary PH was tested with a cohort of 32 patients. True PH status was based on RHC. A diagnosis of PH was established from mPAP >20mmHg, while pre-capillary PH required PCWP ≤ 15mmHg and PVR ≥ 3 Woods Units, and post capillary PH required PCWP > 15mmH and PVR < 3 Woods Units [21]. Patients with both high PVR and PCWP > 15mmHg were classified as combined pre- and post-capillary PH (CpcPH). Subjects with CpcPH were treated as positive for both pre- and post-capillary PH; calculation of PPV — Positive predictive value for Precapillary Pulmonary Hypertension: 86%; positive predictive value = 0.86

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- PVD, Left Heart Disease, Lung Disease: Patients with Pulmonary Vascular Disease (10 subjects), isolated left sided heart failure (10 subjects), and isolated lung disease(10 subjects) will undergo Xe MRI scans with GE-141, Hyperpolarized 129Xenon gas to develop diagnostic criteria for optimizing the sensitivity and specificity of XeMRI for the diagnosis of PVD
  GE-141, Hyperpolarized 129Xenon gas: XeMRI scans will provide 3D images of ventilation and gas exchange. Subjects will inhale HP 129Xe from the dose delivery bags. Then the subject will be moved into the scanner and they will undergo basic 1H localizer and anatomical scans. Once localization is complete, subjects will under-go several MRI scans after inhalation of HPXe
  MRI: Perform MRI scans with administration of GE-141, Hyperpolarized 129Xenon
Arm/Group | PVD, Left Heart Disease, Lung Disease | Pulmonary Vascular Disease
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 0/30 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT03078192/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT03078192/ICF_001.pdf